CLINICAL TRIAL: NCT06493643
Title: Peripheral Perfusion Index as a Predictor of Successful Supraclavicular Brachial Plexus Block in Patients Undergoing Hand Surgeries
Brief Title: Peripheral Perfusion Index as a Predictor of Successful Supraclavicular Brachial Plexus Block
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MS 726/2023
Record Dates: First submitted 2024-05-12; First posted 2024-07-10 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2023-12

CONDITIONS: Perfusion Index
Keywords: Supraclavicular block; Brachial plexus block; Perfusion index ( PI )

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perfusion index at the blocked & unblocked limb: The Perfusion Index was recorded at baseline and at 10, 20, and 30 min after local anaesthetic injection in both the blocked limb and the contralateral unblocked limb using two separate oximeters.
  In every patient , a comparison between the blocked and unblocked limb was performed .
  Interventions: Other: Measurement of perfusion index after supraclavicular brachial plexus block at blocked & unblocked limb

INTERVENTIONS:
Other: Measurement of perfusion index after supraclavicular brachial plexus block at blocked & unblocked limb — The PI (Perfusion Index) was measured using Masimo SET pulse oximetry applied on the index finger. The PI was recorded at baseline and at 10 , 20 , and 30 min after local anaesthetic injection in both the blocked limb and the contralateral unblocked limb using two separate oximeters. The PI ratio was calculated as the ratio between the PI at 10min after injection and the baseline PI. In every patient, a comparison between the blocked and unblocked limb was performed .

SUMMARY:
Aim of the study is to determine the best cut off value for the PI and PI ratio for predication of successful supraclavicular brachial plexus block in young and middle age patients undergoing hand surgeries .

DETAILED DESCRIPTION:
* The supraclavicular nerve block was performed under guidance of a linear transducer (8-14 MHz; Acuson x300; Siemens Healthcare, Seoul, Korea) over the supraclavicular fossa in the coronal oblique plane immediately superior to the midclavicular point. The block was induced in the semi-sitting position, with the head of the patient turned away from the side to be blocked.
* The PI was measured using Masimo SET pulse oximeter, applied on the index finger. The PI was recorded at baseline and at 10, 20, and 30min after local anaesthetic injection in both the blocked limb and the contralateral unblocked limb using two separate oximeters.
* The PI ratio was calculated as the ratio between the PI at 10min after injection and the baseline PI. In every patient, a comparison between the blocked and unblocked limb was performed.
* PI was recorded at baseline and at 10, 20, and 30 min after local anaesthetic injection in both the blocked limb and the contralateral unblocked limb.
* PI ratio was calculated as the ratio between the PI at 10 min after injection and the baseline PI.
* Vital data (Blood pressure, Heart rate, SPO2) was recorded before giving the block and at 10, 20, and 30 min after local anaesthetic injection and at the end of the operation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aging between 15_ 60 years of both sexes.
* Patients undergoing Elective hand Surgeries under successful supraclavicular brachial plexus block anesthesia.
* American Society of Anesthesiologists (ASA) physical status classes I - II.

Exclusion Criteria:

* Patient's refusal of procedure or participation in the study.
* ASA classes III or above.
* Coagulopathy and bleeding disorders.
* Contraindications to supraclavicular brachial plexus block anesthesia such as local infection.
* Hypersensitivity to the study medications.
* Diabetes mellitus.
* Peripheral vascular disease.
* Emergency surgeries.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients undergoing elective hand surgeries at El-demerdash Hospital of Surgery during the study period.
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cut off value for perfusion index ( PI ) for predication of successful supraclavicular brachial plexus block. | Perfusion index (PI) was recorded at baseline and at 10, 20, and 30 minutes after local anaesthetic injection in both the blocked limb and the contralateral unblocked limb.
  Perfusion index (PI) was recorded at baseline and at 10, 20, and 30 minutes after local anaesthetic injection in both the blocked limb and the contralateral unblocked limb.
Cut off value for perfusion index (PI) ratio for predication of successful supraclavicular brachial plexus block. | Perfusion index ( PI ) ratio was recorded at baseline and 10 minutes after local anaesthetic injection
  Perfusion index (PI) ratio was calculated as the ratio between the PI at 10 minutes after injection and the baseline PI.